CLINICAL TRIAL: NCT03410433
Title: Split-mouth Analysis of Different Suture Materials in Periodontal Surgery: Microbiological and Clinical Aspects
Brief Title: Suture Materials: an Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S58697
Record Dates: First submitted 2018-01-18; First posted 2018-01-25 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Suture Materials

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (8):
- Silk 4.0 (Active Comparator): Silk suture
  Interventions: Device: Silk 4.0
- PG910 4.0 (Active Comparator): Vicryl Rapid suture
  Interventions: Device: PG 910 4.0
- PP 4.0 (Experimental): Non-absorbable polypropylene monofilament
  Interventions: Device: PP 4.0
- Silk 5.0 (Active Comparator): Silk suture
  Interventions: Device: Silk 5.0
- PG910 5.0 (Active Comparator): Vicryl suture
  Interventions: Device: PG910 5.0
- PP 5.0 (Experimental): Non-absorbable polypropylene monofilament
  Interventions: Device: PP 5.0
- APG 5.0 (Experimental): Antibacterial Vicryl suture
  Interventions: Device: APG 5.0
- ePTFE 5.0 (Experimental): expanded polytetrafluoroethylene
  Interventions: Device: ePTFE 5.0

INTERVENTIONS:
Device: Silk 4.0 — Silk suture 4.0
  Arms: Silk 4.0
Device: PG 910 4.0 — PG 910 4.0
  Arms: PG910 4.0
Device: PP 4.0 — PP 4.0
  Arms: PP 4.0
Device: Silk 5.0 — Silk 5.0
  Arms: Silk 5.0
Device: PG910 5.0 — PG910 5.0
  Arms: PG910 5.0
Device: PP 5.0 — PP 5.0
  Arms: PP 5.0
Device: APG 5.0 — APG 5.0
  Arms: APG 5.0
Device: ePTFE 5.0 — ePTFE 5.0
  Arms: ePTFE 5.0

SUMMARY:
Background: Many factors play a role when selecting an appropriate suture for optimal soft tissue healing in oral surgery. Moreover, the oral cavity has its specific challenges: it is an aqueous environment in which biofilm formation takes place on all surfaces. Therefore, oral surgery has specific demands for suture materials.

Aim: The primary objective of this study was to compare the bacterial load on different suture materials. The secondary objective was to determine the impact of suture material on decubitus.

Material & methods: This prospective experimental study with a 'split-mouth' design enrolled 36 patients requiring oral surgery. Five different suture materials were compared regarding their microbiological load and decubitus at the suture removal. Bacterial accumulation on the same 5 suture materials was also tested in an in vitro biofilm model.

ELIGIBILITY:
Inclusion Criteria:

* 36 patients
* in need for periodontal surgery
* patients in good general health
* able to sign IC form

Exclusion Criteria:

* patients that were deemed unlikely to comply with the study protocol, as judged by the examiner
* patients who had a present alcohol and/or drug abuse

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Accumulation of soft deposits | 7 to 14 days
  Accumulation of soft deposits on each suture material was assessed visually as being present or absent before removing the knots.

SECONDARY OUTCOMES:
Area of inflammation | 7 to 14 days
  Clinical photographs were taken, calibrated with a ruler of 0.5 mm accuracy as is illustrated in Figure 2, before and after suture removal in both parts of the clinical study. Subsequently, the area of inflammation surrounding the sutures was measured by two separate examiners using the image-analysis program, Image J® (NIH, Bethesda, Maryland, USA).
Microbial deposits on the sutures | 7 to 14 days
  The composition of the microbial deposits on the suture materials was examined with qPCR.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Quirynen, Study Director — KU Leuven

IPD SHARING:
Plan to Share IPD: No